CLINICAL TRIAL: NCT06381635
Title: Synergistic Effect of Aloe Vera Gel and Manuka Honey on Radiation Induced Oral Mucositis in Head and Neck Cancer Patients: Randomized Controlled Clinical Trial
Brief Title: Effect of Aloe Vera Gel and Manuka Honey on Radiation Induced Oral Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FD-BUE-REC: IRB000124920
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Radiation Mucositis
MeSH Terms: interventions — Aloe vera gel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): patients will be given 20 mL of Manuka honey with aloe vera gel, 15 min before and after the radiotherapy. They were instructed to swallow slowly to smear the layer of honey on the oral and pharyngeal mucosa. Patients were also advised to take 20 mL of Manuka honey before sleeping in the night. This treatment protocol was followed from day 1 of radiation till 6 weeks.
  Interventions: Dietary Supplement: Manuka honey mixed with aloe vera gel
- Control group (Placebo Comparator): patients will be given 20 mL of 0.9% of saline 15 min before and after radiotherapy [54]. They will be advised to rinse saline. They will be instructed to keep saline for at least 5 min duration and then to spit it out. They will be advised to rinse 20 mL of saline in the same manner before sleeping. This treatment protocol was followed from day 1 of radiation till 6 weeks.
  Interventions: Dietary Supplement: Manuka honey mixed with aloe vera gel

INTERVENTIONS:
Dietary Supplement: Manuka honey mixed with aloe vera gel — a mix gel of manuka honey and with aloe vera honey (1:1) mixed in water bath to get a homogenous mix is then packed in unmarked bottles.

SUMMARY:
The goal of this [ type of study: Clinical trial] is to test effectiveness of Aloe Vera Gel and Manuka Honey in management of Radiation Induced Mucositis in head and neck cancer patients.

The main question [s] ] is to [ learn about, test, compare etc.] it aims to answer are:

1. Is Aloe Vera Gel and Manuka Honey effective in management of Radiation Induced Mucositis?
2. Does Aloe Vera Gel and Manuka Honey affect the level of TGFβ1 and EGF in saliva of patients with radiation induced mucositis? participants will be asked to apply Aloe Vera Gel and Manuka Honey or saline three times daily during radiotherapy and 6 months after radiotherapy.

DETAILED DESCRIPTION:
Head and neck cancer is the eighth common type among all cancer types all over the world [1] The treatment comprises surgery, radiotherapy, chemotherapy or a combination escorted by restoration therapy, and social support [2] Radiotherapy leads to irreversible loss of the reproductive integrity, the cell cycle necessary for cell growth, apoptosis, and necrosis of cancer cells [3] Conventional fraction size ranges from 1.8 to 3 Grays (Gy) per fraction over 4-6 weeks [4] The accumulative dose of radiation for the primary treatment of head and neck cancer treatment is 60-70 Gy, depending on the irradiation of the tumor [5].

Radiation affects malignant cells and is also absorbed by the oral mucosa and gastrointestinal mucosa, especially in rapidly dividing cells [6] Oral mucositis is the most frequent, distressing, painful, clinical side effect of radiotherapy [7] It is defined as an inflammatory lesion of oral mucosa resulting from the cancer therapy typically manifesting as atrophy, swelling, erythema, ulceration, and pseudomembrane formation [8,9] It is described in five overlapping stages: initiation, upregulation, message generation, ulceration, and healing [9,10].

Radiation-induced oral mucositis shows hyperkeratosis of the oral mucosa after the dose of 10-20 Gy [6,8] Erythema is the first clinical sign seen on the oral mucosa, and severity of mucositis reaches at a dose of 30 Gy. After the completion of radiotherapy, the symptoms abate in 2-6 weeks [11,12] Effective management of oral mucositis is very important [13,14].

Honey is an important traditional medicine and prophylactic agent that has numerous beneficial health properties including its ability to facilitate healing.[15,16] Honey helps in the reduction of ulceration and inflammation of the biological process of mucositis.[17,18] Honey has been used to manage burns, oral infections, surgical wounds, and pressure wounds.[19,20]. Honey was applied to the oral mucosa of patients undergoing radiotherapy which is beneficial in limiting the severity of oral mucositis. Honey is a natural product with rich nutritional properties that is economical and a pleasant agent for managing mucositis [21].

Manuka honey is a monofloral honey, produced from the nectar of flowers of Manuka tree. This variety is produced from the Apis mellifera honey bees, using New Zealand Manuka plants producing specific floral-variety named as Leptospermum scoparium [22]. Manuka honey is usually rated using a classification system known as the Unique Manuka Factor (UMF), which reflects the equivalent concentration of phenol (%, w/v) required to produce the same antibacterial activity as honey.

The composition of Manuka honey consists of carbohydrates, minerals, proteins, fatty acids, phenolic and flavonoid compounds. Although such compounds are found in other types of honey, other unique features also occur in Manuka honey, such as an unusually high level of methylglyoxal (MGO) formed from dihydroxyacetone (DHA) which correlates with antibacterial activity [23, 24]. Kato et al. also noted the occurrence of methyl syringate glycoside (leptosperin) as a unique maker for Manuka honey authentication [25]. Interestingly, the UMF rating of Manuka honey strongly correlates with MGO equivalence and antibacterial activity but the relation is not wholly understood [26]. In addition to antibacterial activity [22, 26], UMF honey has the ability to stimulate macrophages through Apalbumin 1 protein to release mediators such as TNF-α, IL-1β and IL-6, which are needed for reducing microbial infections and helping in tissue healing [27]. Manuka honey shows antioxidant and anticancer properties, which are considered due to its constituents-phytochemicals working as active bio-compounds [28, 29].

Aloe Vera (AV) is a cactus-like plant that grows readily in hot, dry climates. It belongs to the Liliacea family, of which there are about 360 species. Only two species are grown commercially: Aloe barbadensis Miller and Aloe aborescens. The parenchymatous cells in the fresh leaves of aloe vera secrete colorless mucilaginous gel (i.e., Aloe vera gel) that contains 98-99% water and 1-2% active compounds [30, 31] Aloe vera gel has various pharmacological actions like antibacterial, antifungal, anti-inflammatory, antioxidant, antitumour, hypoglycaemic properties and immune boosting. Therefore it is used traditionally as nutritional drinks, moisturizer, healing agent in cosmetics, diabetic patients, sun burn, wounds and digestive tract disorders, there is no adverse effect [32].

Aloe vera gel had also been used in dentistry and showed good results. It had been used for treatment of over extraction socket and endodontic medicament. Various dentifrices also contains Aloe vera gel as its constituent because of its medicinal property [33-34]. Studies have demonstrated that aloe vera has an important therapeutic uses in the management of oral lesions such as oral lichen planus, oral submucous fibrosis, radiation induced mucositis, burning mouth syndrome, xerostomia, recurrent apthous ulcers [31].

Transforming growth factor-β (TGF-β) is a family of related proteins that regulate many cellular processes including growth, differentiation, extracellular matrix formation and immunosuppression [35]. TGF-β protein is produced by nearly all normal cells and functions through a complex cell surface receptor system [36].

The three mammalian isoforms of TGF-β (TGF-βs 1, 2, and 3) have similar but distinct functions and are approximately 70% identical in amino acid sequence. Transforming growth factor-β (TGF-β) proteins and their antagonists have entered clinical trials. These multi-functional regulators of cell growth and differentiation induce extracellular matrix proteins and suppress the immune system making TGF-βs useful in treatment of wounds with impaired healing, mucositis, fractures, ischemia-reperfusion injuries, and autoimmune disease. In diseases such as keloids, glomerulonephritis and pulmonary fibrosis, excessive expression of TGF-β has been implicated as being responsible for accumulation of detrimental scar tissue. In these conditions, agents that block TGF-β have prevented or reversed disease. Similarly, in carcinogenesis, blocking TGF-β activity may be valuable in stimulating an immune response towards metastasis. As these blocking agents receive approval, we will likely have new therapies for previously recalcitrant diseases [37]. It has been stated that transforming growth factor-β3 (TGF-β3) negatively regulates epithelial cell proliferation and reduces the incidence of oral mucositis [38].

A great number of growth factors and cytokines are involved in the wound site [39]. Of the growth factors, basic fibroblast growth factor (bFGF), transforming growth factor (TGF-b), and platelet-derived growth factor (PDGF) are anti-inflammatory and the most important in the wound healing process [40]. The bFGF (FGF-2) is a member of the FGF's family and has been shown in several studies to be an essential growth factor for fibroblast and vascular endothelial cell [41]. bFGF is increased in acute wound healing and plays a role in granulation tissue formation, re-epithelization, and tissue remodeling [42]. Although clinical studies have shown that bFGF was not successful in the treatment of diabetic foot ulcers, topical bFGF application has been found to increase the healing of burns and venous ulcers [43, 44, 45]. Moreover, TGF-β and PDGF are both crucial for inflammation, granulation, angiogenesis, connective tissue regeneration, re-epithelization, and remodeling which stimulate macrophages by increasing the secretion of other growth factors [43, 46]. They stimulate collagen production, affect matrix formation, and inhibit metalloproteinase (MMP) activity, which degrades collagen deposition. Levels of PDGF, TGF-β, and FGF are decreased in chronic wounds.

Epidermal growth factor (EGF), first discovered in the submaxillary gland of a rat in 1962, comprises a single-chain polypeptide containing 53 amino acids [47, 48]. EGF was later discovered in various normal tissues and body fluids, including the skin, mucosa, tears, cornea, saliva, milk, semen, and fluids secreted by the duodenal glands [49, 50]. EGF helps maintain tissue homeostasis by regulating epithelial cell proliferation, growth, and migration. It also induces angiogenesis, which provides nutritional support for tissues. Thus, EGF plays an important role in wound healing and tissue generation and may be useful in the treatment of radiation-induced oral mucositis [51, 52].

ELIGIBILITY:
Inclusion Criteria:

* a) Patients with a confirmed histologic diagnosis of H&N malignancy who are referred to non-palliative radiotherapy in the oral cavity.

  b) Patient who is receiving radiation therapy with IMRT or 3D techniques. c) Patients received 50-70 Gy of total radiation at the rate of 2 Gy/fraction daily and 5 fractions/week.

  d) Patient who received concurrent chemotherapy with radiotherapy e) Presence of Oral Mucositis f) Age 20-70 years old g) Willing to participate in the study. h) Able to complete the study assessments.

Exclusion Criteria:

* a) Have a confirmed or medically treated diabetes mellitus b) Radiotherapy within the last 6 months prior to this study c) Vulnerable patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from World Health Organization Oral Toxicity Scale Grading of Oral Mucositis | Three points: -"baseline which is at the starting of radiotherapy", -"the second of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline, while the end point is after six months of radiotherapy.
  World Health Organization Oral Toxicity Scale Grading of Oral Mucositis ranges from "1,2,3,4) the grade1 me

SECONDARY OUTCOMES:
the level of salivary transforming growth factor beta 1 | Two points: -"baseline which is at the second week of radiotherapy" while -"the end of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline.
  salivary level of transforming growth factor beta 1 assessment using enzyme linked immune assay may range from 10-4000ng/L
the level of salivary Epidermal Growth factor (EGF) | Two points: -"baseline which is at the second week of radiotherapy" while -"the end of the radiotherapy is at seventh week of the radiotherapy or 4-5 weeks from baseline.
  salivary level of Epidermal Growth factor assessment using enzyme linked immune assay may range from 3.9-250 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Fatma E. Hassanein, PHD, Study Director — lecturer
Locations (2):
- Egypt (2):
  - ain shams University, Cairo
  - Fatma E.Sayed, Cairo

IPD SHARING:
Plan to Share IPD: No